CLINICAL TRIAL: NCT00763607
Title: Retrospective Study Evaluating IGF1R And p95HER2 as Prognostic Factors in Radically Resected Non Small Cell Lung Cancer
Brief Title: Retrospective Study Evaluating IGF1R And p95HER2 as Prognostic Factors in Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-02/2007
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorescent Antibody Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Paraffine embedded tumor sections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Radically resected Non small cell lung cancer patients in stage I-III
  Interventions: Genetic: Protein expression by immunohistochemistry and immunofluorescence

INTERVENTIONS:
Genetic: Protein expression by immunohistochemistry and immunofluorescence — Protein expression by immunohistochemistry and immunofluorescence

SUMMARY:
Aim of the study is to evaluated the role of IGF1R and p95HER2 on prognosis in radically resected non small cell lung cancer patients

The primary objective is to correlate the expression of IGF1R and p95HER2 with survival.

ELIGIBILITY:
Inclusion Criteria:

* Radically resected non small cell lung cancer patients with tumor tissue available

Exclusion Criteria:

* Tumor tissue not available
* Clinical data not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radically resected non small cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Association of different biomarkers with survival | At the end of enrollment

SECONDARY OUTCOMES:
Association of a specific biomarker with patient's characteristics | At the end of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milan, Italy